CLINICAL TRIAL: NCT00243620
Title: State-of-the Art Treatment of Chronic Leg Ulcers: a Randomised Controlled Trial Comparing Vacuum Assisted Closure (V.A.C.®) With Modern Wound Dressings
Brief Title: A Randomised Controlled Trial Comparing Vacuum Assisted Closure (V.A.C.®) With Modern Wound Dressings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: KCI medical B.V (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB/jd/01.259
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2001-05

CONDITIONS: Leg Ulcer
Keywords: Chronic leg ulcers; wound healing; wound care; Vacuum Assisted Closure; topical negative Pressure
MeSH Terms: conditions — Leg Ulcer

INTERVENTIONS:
Device: Vacuum therapy (device)

SUMMARY:
Current treatment modalities for chronic leg ulcers are time consuming, expensive, and only moderately successful. Recent data suggest that creating a sub-atmospheric pressure by Vacuum Assisted Closure (V.A.C.®) therapy supports the wound healing process. Here, we studied the efficacy of V.A.C.® in the treatment of chronic leg ulcers prospectively.

DETAILED DESCRIPTION:
PROTOCOL

I. INTRODUCTION:

In the last 25 years we have entered an area where patients are living longer with more complex systemic pathology. The number of patients with chronic non-healing wounds continues to increase, despite many recent advances in the basic science of wound healing.

Although, the chronic leg ulcers approximately affect 1 % of the adult population of developed countries and chronic wound care consumes 1-2% of the health care budgets of European countries. It is still probably true to say that leg ulcer disease is not sufficiently recognised as a problem either by the population at large or by the medical community. Recent socio-economic and quality of life data showed the importance of this long-neglected health care problem.

In recent years, many new wound care products were developed. We have learned that a moist wound bed, without maceration of wound borders, gives faster wound healing. So, wound care products need a high absorption capacity and at the same time, they need to create a moist wound climate. However, many of these new wound care products resulted in divergent results. Complications are described like enlargement of the wounds, maceration, infections, sepsis and loss of grafts. These results in delayed hospitalisation and increased costs.

In 1989 Prof. Argenta and Dr. Morykwas developed a sub-atmospheric pressure technique: " Vacuum Assisted Closure". This technique was introduced to our hospital by the department of surgery in the treatment of large complicated surgical wounds.

We are employing this new technique at our department of dermatology in treating lower leg ulcers since 1997, by placing a foam dressing into the wound, seal it with tape and applying a sub-atmospheric pressure to the wound.

The meaning of Vacuum Assisted Closure is, first to clean the ulcer in a quick and non-invasive way until a vital red wound is produced (first stage). When a wound is too big to close primarily, secondary surgery is needed. By using the V.A.C.-technique in combination with transplantation, the skin grafts will be supported in adhering to the wound surface (second stage).

Before the PVA (Polyvinylalcohol) or PU (Polyurethane ether) foam is placed into the wound, the border has to be protected by hydrocolloïd foam, which will be trimmed to the appropriate size and geometry for each individual wound. After that, The PVA or PU foam can be placed into the wound defect. We employed especially a reticulated polyvinyl alcohol dressing with a pore size of 400-600 h-meters depending of the appearance of the wound bed. The Polyurethane ether foams were often used in the past. The PVA or PU foams are embedded with a non-collapsible evacuation tube, having side ports that allow communication of the lumen to the space of the reticulated foam. In large wounds, multiple foams may be placed in close contact to one another. The surface of the foam dressing is covered by an adhesive drape, extending 5 cm, beyond the hydrocolloid dressings. The proximal end of the evacuation tube leads to a collection canister localised on the V.A.C. pump into which the wound fluid will be drawn when a permanent sub-atmospheric pressure is applied. So an open wound is now converted to a controlled closed wound.

First a permanent subatmospheric pressure was applied to the chronic ulcus cruris until a vital red wound was produced (first stage). Subsequently, these ulcers were treated by a combination of transplantation and vacuum sealing to support the skin grafts (the second stage). The therapy was monitored weekly.

The V.A.C. is the first active, non-invasive wound care product, used by a secure local regulated sub-atmospheric pressure technique.

The exact mechanisms to explain this treatment are not known yet. Researches by Prof. Argenta et al. postulated that interrelated factors are the basis for the success of the technique. These factors can be devised in 3 subgroups: (1) Removing, (2) Improving, (2) Reducing

1. Tissues surrounding the chronic wounds are characterised by localised collection of interstitial or third-space fluid. This collection of third-space fluid contains factors which inhibits or suppresses mitosis, protein synthesis and fibroblasts collagen synthesis. An active withdrawal of this fluid removes the excess of third space wound fluid and its inhibitory factors. The active withdrawal also results in the removing of wound debris.
2. The collection of third space fluid mechanically comprises the micro-vascularisation and lymphatic system. By removing the third space fluid and its inhibitory factors, this result in increased vascularisation, reduced venous afterload and an increased delivery of oxygen and nutrients as well. These changes improve the rate of granulation formation and the concentration of growth factors. An additional mechanism of the V.A.C. is the mechanical stimulation of cells migration by tensile forces placed on the surrounding tissues.
3. Besides reducing of third space fluid, we know that successful wound healing correlates with bacterial counts of less than 100 000 organism per gram of tissue.

Bacterial counts of human wounds treated by V.A.C. have demonstrated a significant decrease after 3-4 days usually until less than 1000 per gram of tissue. Last but not least, the V.A.C. technique also reduces the infection chances, because the creation of a controlled closed wound.

Recently socio-economic and quality of life evaluation showed the impact of this long-neglected health care problem. Phillips et al shows a strong correlation between time spent on ulcer care and feelings of anger and the quality of life. Besides that, there is no doubt that ulcer care consumes a substantial proportion of the health care budgets. The retrospective results of V.A.C. therapy compared to the conventional therapy showed a reduction up tot 39% in hospitalisation time. These outcomes may be result in a better quality of life and a reduction of the health care costs.

Summarised V.A.C. treatment has a positive effect to wound cleaning and increases the survival chance of transplanted skin, which will minimise hospitalisation time and costs, compared to the conventional wound care techniques. It must be emphasised that the Vacuum-assisted Closure technique was developed as an adjunct to wound care. It is not meant to, and will never, replace surgical procedures. Despite the positive effects, this method needs more and further investigation.

A randomised, prospective, comparative cost/ effect balance and quality of life investigation will be starting soon in co-operation with Prof. H.A.M. Neumann (University Hospital Maastricht), comparing the V.A.C. treatment versus conventional therapy.

II. AIMS OF THIS MULTI-CENTRE STUDY:

To demonstrate V.A.C. therapy is a more quick and cheap option in the treatment of chronic arteriolosclerotic, chronic venous en combined venous /arterial leg ulcers.

III. PATIENTS AND METHODS:

3.1 Patients: The study is conducted in the departments of Dermatology at the University Hospital Maastricht and the Atrium Medical Centre Heerlen. All patients in which extensive ambulatory treatment in an out-patient-clinic according to the Scottish Intercollegiate Guideline Network (SIGN) had failed and who are hospitalized due to chronic venous (venous insufficiency of the deep or superficial system without an arterial incompetence), combined venous/arterial (venous insufficiency of the deep or superficial system with an ankle/brachial index of 0·60 - 0·85) or arteriolosclerotic (Martorell's ulcer) leg ulcers, are evaluated for eligibility in this study.

3.2 Methods: Patients are randomly assigned to the VAC® therapy group or to the control group (conventional wound care) by a computer program using random permuted blocks of 8. Randomisation was carried out within 3 strata, one for each ulcer type: venous, combined venous/arterial, and arteriolosclerotic ulcers, respectively. Treatment allocation occurred through telephone calls to the coordinating centre.

In both study groups and both study centres an initial necrotectomy was performed by sharp debridement of slough and nonviable tissue.

I.Vacuum Assisted Closure-techniques:

Before the PVA (Polyvinylalcohol) or PU (Polyurethane ether) foam is placed into the wound, the border has to be protected by a hydrocolloïd foam, which will be trimmed to the appropriate size and geometry for each individual wound. After that, The PVA or PU foam can be placed into the wound defect. We employed especially a reticulated polyvinyl alcohol dressing with a pore size of 400-600 h-meters depending of the appearance of the wound bed. The Polyurethane ether foams were often used in the past. The PVA or PU foams are embedded with a non-collapsible evacuation tube, having side ports that allow communication of the lumen to the space of the reticulated foam. In large wounds, multiple foams may be placed in close contact to one another. The surface of the foam dressing is covered by an adhesive drape, extending 5 cm, beyond the hydrocolloid dressings. The proximal end of the evacuation tube leads to a collection canister localised on the V.A.C. pump into which the wound fluid will be drawn when a permanent sub-atmospheric pressure is applied. So an open wound is now converted to a controlled closed wound.

The meaning of Vacuum Assisted Closure is, first to clean the ulcer in a quick and non-invasive way until a vital red wound is produced (first stage). When a wound is too big to close primarily, secondary surgery is needed. By using the V.A.C.-technique in combination with transplantation, the skin grafts (punch grafts) will be supported in adhering to the wound surface (second stage). Once all skin grafts are well adhered, the V.A.C. therapy can be stopped. Until 100% wound-closing patients will be hospitalised by compression and local therapy.

Thereafter ambulant therapy (compression and local therapy) will be continued until complete wound healing. Also therapy will be controlled once a week.

II.The conventional wound care techniques (control group):

Patients assigned to standard wound care receive daily local wound care according to the SIGN guideline and a multiple-layer compression bandage (Smith and Nephew, Hoofddorp, the Netherlands) until complete healing. Four basic types of commercially available wound dressings will be used in this study including hydrogels (Johnson&Johnson, Amersfoort, the Netherlands), alginates (Hartmann, Nijmegen, the Netherlands), hydrocolloids (Smith and Nephew, Hoofddorp, the Netherlands), and films (Hartmann, Nijmegen, the Netherlands). The choice of dressing most depended on the ulcer type, the amount of exsudate and the physician's preference. Once 100% granulation was achieved, these patients also received punch skin-graft transplantation in combination with topical therapy.

In both treatment groups, only toilet and basic hygiene mobility was permitted during the wound bed preparation and transplantation stage. After complete wound healing, community-grade elastic support stockings class 2 (Medi, Breda or Varodem, Horn; the Netherlands) or 3 (Varodem, Horn; the Netherlands) were prescribed depending on the underlying pathology.

3.3 Punch transplantation procedure The transplants will be taken of the upper-leg by placing first a 'field-block' local anaesthetic (lidocaine 2% in NaCl). Epidermal grafts will be created using a biopsy corer of 4 mm). The size of the field-block depends of the ulcer size.

3.4 Evaluation criteria Because masking the interventions is not possible, patients will be reviewed clinically by the same independent research physician and consultant dermatologist twice a week until the ulcer is healed: description of the wound defect, surrounding tissue, tracing the ulcer and taking a picture (Enclosure III), time investment forms (nurse and MD) (Enclosure IV), evaluation of the used materials (Enclosure IV), evaluation of the V.A.C. therapy and noting complications (Enclosure IV) and the quality of life evaluation of the patient (Enclosure II). Using codes will anonymise all the patient information.

3.5 Selection criteria:

1. Patient groups (V.A.C.; n=30 / Conventional techniques; n=30):

   I.chronic venous leg ulcer II. chronic combined venous /arterial leg ulcer III. chronic arteriolosclerotic leg ulcer
2. Sex : either sex
3. Inclusion criteria:

   a)patient with a chronic leg ulcer (> 6 months) without healing signs and satisfies to one or more criteria:
   * Venous (venous insufficiency of the deep or superficial system without an arterial incompetence)
   * Combined venous/arterial (venous insufficiency of the deep or superficial system with an ankle/brachial index of 0·60 - 0·85)
   * Arteriolosclerotic (Martorell's ulcer) leg ulcers (diagnose made by anamnesis, clinical signs, exclusions of differential diagnosis's, venous/ arterial duplex shows no signs of obstruction or major venous insufficiency, histology)
4. Exclusion criteria:

1) ulcer duration shorter than 6 months 2) age > 85 years 3) use of immune suppressive medication 4) known type IV allergies against ingredients of the wound care products 5) insulin-dependent diabetes mellitus type I 6) severe peripheral arterial disease (ankle/brachial index <0·60) 7) vasculitic ulcers 8) neoplastic ulcers. In patients presenting with multiple ulcerations, the clinically most severe ulcer was included in the study whereas the other ulcers were treated conventionally.

3.6 Informed Consent :

Written informed consent will be obtained from all patients (volunteers). The investigator will explain the nature of this study and its purpose, risks and duration.

Patients (volunteers) will advised that they are free to participate in, or to withdraw from, the study at any time without prejudice to the doctor-patient relationship. The medical care provided will not be affected or refusal to participate in this study.

This protocol will be submitted to the appropriate institutional Ethical Committee and their approval obtained in writing will be awaited before starting the study.

3.7 Randomisation:

All volunteers first will underwent a complete intake. When the volunteer satisfy the inclusion- and exclusion criteria, this multi-centre trial the randomisation procedure will be carried out by the clinician being in contact with a central registration office, by telephone. An independent person will use a computer program, which determine the therapy (V.A.C. or Conventional therapy) by serial numbers. This centralisation helps the correct implementation of each step and ensures that someone has an overview of how the trial is going. Before randomisation, stratification into the ulcer type (3 strata: venous, combined venous/ arterial and arteriolosclerotic ulcers) is needed. Using codes will anonymise all patient information.

Data from a retrospective study showed that the mean duration of the preparation period was 24 days in conventional wound care (SD 11) versus 12 days in VAC® therapy (SD 5). In order to detect a minimal difference of 10 days in preparation time with a power of 80% (α=5%) the number of patients required in each treatment-group was 30, as derived from sample-size calculations.

3.8 Masking: Because masking the interventions is not possible, patients were reviewed clinically by the same independent research physician and consultant dermatologist twice a week until the ulcer had healed. Thereafter, patients were prospectively followed up by one and the same research physician at three months, six months and one year after discharge. All participating clinicians completed standardised case record forms and checklists during their control visits, treatments and follow-ups.

Decisions made during the treatment (V.A.C. and conventional therapy) are based on simple and objective standards:

* Yellow debris and a necrotic tissue is bad climate for skin grafts.
* Only a red, vital granulated wound bed causes a successful transplantation
* Once all skin grafts are well adhered, the V.A.C. therapy can be stopped.
* 100% epithelialisation (wound closure) This approach seems to be authorised, because scientific investigations showed these kinds of judgements are apparent equally objective compared to other judgement methods (thesis of Dr. Mekkes; Amsterdam). To have an external control, every intervention will be photograph.

3.9 outcome results:

Primary endpoints:

Time-to-complete-healing: i.e. the period between initial preparation of the wound and 100% epithelialisation with the primary endpoint being time-to-complete-healing.

Secondary endpoints:

1. duration of the wound-bed preparation stage
2. percentage of leg ulcer recurrences within one year (i.e. an epithelial breakdown anywhere along or within the index ulcer region)
3. skin-graft survival, where applicable (i.e. percentage of successfully adhered skin grafts after 4 days of complete bed rest and compression or VAC® treatment) Furthermore, we compared between both experimental groups i) the quality of life, ii) pain scores, iii) the total time needed for wound care until complete wound closure, and iv) the costs per ulcer.

3.10 Follow-up: Patients are followed up by one and the same research physician at three months, six months and one year after discharge.

3.11 Statistical analysis: All data will be analysed using the SPSS 11.0 software package and the results are analysed on an intention-to-treat basis. Time-to-complete-healing, duration of wound-bed preparation, and recurrence rates are compared using the Kaplan-Meier survival analysis. The log rank test is used to test for statistically significant differences between both groups. Multivariate Cox's regression analysis is used to adjust for imbalances in the baseline distribution of relevant prognostic factors. The regression coefficient, expresses the independent contribution of potential determinants to duration of cleaning and wound-healing. Hazard ratios and their 95% confidence intervals (95% CI) are presented. A p-value of less than 0·05 was considered to be statistically significant.

Percentages are compared by the chi-square test and continuous variables are compared using the independent samples t-test (for normally distributed variables) and the two-independent sample test (for non-normally distributed variables).

LITERATURE:

1. C.Jane Morell, Stephen J Walters, Simon Dixon at al., Cost effectiveness of community leg ulcers clinics: randomised controlled trial. BMJ 1998; vol. 316: 1487-1491
2. C.B. Ruckley, ChM FRCSE, Socioeconomic Impact of chronic venous insufficiency and leg ulcers. Angiology 1997; vol. 48: 67-69
3. Bradley M, Cullum N, Nelson EA, Petticrew M, Sheldon T, Togerson D. Systemic reviews of wound care management: Dressings and topical agents used in the healing of chronic wounds. Health Technology Assessment 1999;3(17 Pt 2):1-78.
4. Simon DA, MCCollum CN. Approaches to venous leg ulcer care within the community: compression, pinch skin grafts and simple venous surgery.

   Ostomy Wound Manage. 1996 Mar;42(2):34-8, 40. PMID: 8703294; UI: 96340071
5. Louis C. Argenta, M.J. Morykwas, Vacuum-Assisted Closure: A new method for wound control and treatment: Clinical Experience. Annals of Plastic Surgery 1997; vol. 38: 562-576
6. M.J. Morykwas, L.C. Argenta, E.I. Shelton-Brown, W. McGuirt, Vacuum-Assisted Closure: A new method for wound control and treatment: Animal studies and basic foundation. Annals of Plastic Surgery 1997; 38, no 6: 552-561
7. M.J. Morykwas, L.C. Argenta, Nonsurgical modalities to enhance healing and care of soft tissue wounds. Journal of the Southern Orthopaedic Association 1997; vol. 6, no 4: 279-288
8. J.D.D. Vuerstaek, J.C.M.J. Veraart, J.Wuite, A.M.J. van der Kley, Een nieuw concept voor actieve wondbehandeling; Vacuum Assisted Closure (V.A.C.). Scripta Phlebologica 1999; vol. 7, 55-57
9. Falanga V, Growth factors and chronic wounds: the need to understand the microenvironment. J Dermatology 1992; 19: 667-672
10. Bucalo B, Eaglstein WH, Falanga V, Inhibition of cell proliferation by chronicle wound fluid. Wound Rep Regen 1993; 1: 181-186
11. Wyocki AB, Staiano-Coico L. Grinnell F. Wound fluid from chronic leg ulcers contains elevated levels of metaloproteinases MM-2 and MMP-9, J Invest Dermatol 1993; 101: 64-68
12. Thoma R. Ueber die histomechanik des gefassystems und die pathogenese der angioskleroose. Virchows Arch F, Path Anat 1911; 204:1-74
13. Ilizarov GA, The tension-stress effects on the genesis and growth of tissues. Part I, Clin Orthop Rel Res 1989; 238: 249-281
14. Ilizarov GA, The tension-stress effects on the genesis and growth of tissues. Part II, Clin Orthop Rel Res 1989; 239: 263-285
15. Daltrey DC, Rhodes B., Chattwood JG, Investigation into the microbial flora of healing and non-healing decubitus ulcers. J Clin Path 1981; 34: 701-705
16. Urschel JD, SCOTT PG, Williams HTG, The effect of mechanical stress on soft and hard tissue repair a review. Br J Plast Surg 1988; 41: 182-186

ELIGIBILITY:
Inclusion Criteria:

patient with a chronic leg ulcer (> 6 months) without healing signs and satisfies to one or more criteria:

* Venous (venous insufficiency of the deep or superficial system without an arterial incompetence)
* Combined venous/arterial (venous insufficiency of the deep or superficial system with an ankle/brachial index of 0·60 - 0·85)
* Arteriolosclerotic (Martorell's ulcer) leg ulcers (diagnose made by anamnesis, clinical signs, exclusions of differential diagnosis's, venous/ arterial duplex shows no signs of obstruction or major venous insufficiency, histology)

Exclusion Criteria:

1. ulcer duration shorter than 6 months
2. age > 85 years
3. use of immune suppressive medication
4. known type IV allergies against ingredients of the wound care products
5. insulin-dependent diabetes mellitus type I
6. severe peripheral arterial disease (ankle/brachial index <0·60)
7. vasculitic ulcers
8. neoplastic ulcers.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2001-05; Study Completion 2004-05

PRIMARY OUTCOMES:
Time-to-complete-healing: i.e. the period between initial preparation of the wound and 100% epithelialisation with the primary endpoint being time-to-complete-healing.

SECONDARY OUTCOMES:
1)duration of the wound-bed preparation stage
2)percentage of leg ulcer recurrences within one year (i.e. an epithelial breakdown anywhere along or within the index ulcer region)
3)skin-graft survival, where applicable (i.e. percentage of successfully adhered skin grafts after 4 days of complete bed rest and compression or VAC® treatment)
4) the quality of life
5) pain scores
6) the total time needed for wound care until complete wound closure
7) the costs per ulcer.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Vuerstaek, MD, Principal Investigator — Department of dermatology, UniversityHospital Maastricht; Peter Steijlen, Prof., Study Chair — Department of dermatology, University Hospital Maastricht
Locations (1):
- MUMC, Nederland, Zuid-Limburg, Netherlands